CLINICAL TRIAL: NCT03584516
Title: GRAVITAS-309: A Phase 2/3 Study of Itacitinib and Corticosteroids as Initial Treatment for Chronic Graft-Versus-Host Disease
Brief Title: GRAVITAS-309: Itacitinib and Corticosteroids as Initial Treatment for Chronic Graft-Versus-Host Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to insufficient efficacy to support moving into Part 2 of the study; there were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 39110-309; 2018-001606-29 (EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Graft-versus-host-disease; itacitinib; Janus kinase inhibitor; corticosteroids
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — itacitinib; INCB039110; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisone

STUDY DESIGN:
Intervention Model Description: In Part 2 of the study, participants in the placebo group will be allowed to cross over to the experimental group after completion of the primary analysis.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 : Dose determination of itacitinib (Experimental): itacitinib administered in combination with corticosteroids.
  Interventions: Drug: Itacitinib; Drug: Methylprednisolone; Drug: Prednisone
- Part 1 : Dose expansion of itacitinib (Experimental): itacitinib administered in combination with corticosteroids or corticosteroids alone.
  Interventions: Drug: Itacitinib; Drug: Placebo; Drug: Methylprednisolone; Drug: Prednisone
- Part 2 : itacitinib recommended dose from part 1 (Placebo Comparator): itacitinib or placebo administered in combination with corticosteroids
  Interventions: Drug: Itacitinib; Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Itacitinib — In Part 1dose determination participants will receive itacitinib administered orally once daily at the protocol-defined dose according to cohort enrollment. In Part 1 expansion, participants will receive either itacitinib administered orally either once daily or twice a day or corticosteroid alone based on the assigned treatment regimen according to cohort enrollment. In Part 2, participants will receive the recommended dose from Part 1 expansion.
  Other Names: INCB039110
Drug: Placebo — In Part 2, participants will receive matching placebo.
  Arms: Part 1 : Dose expansion of itacitinib
Drug: Methylprednisolone — Administered in Parts 1 and 2 as background reference therapy at a dose level that is commensurate with institutional guidelines based on organ involvement and severity of disease.
  Other Names: Medrol, Medrol Dosepak, Solu-Medrol
Drug: Prednisone — Administered in Parts 1 and 2 as background reference therapy at a dose level that is commensurate with institutional guidelines based on organ involvement and severity of disease.
  Other Names: Deltasone, Prednicot, predniSONE Intensol, Rayos, Sterapred, Sterapred DS

SUMMARY:
The purpose of this study is to assess the efficacy and safety of itacitinib in combination with corticosteroids as first-line treatment for moderate or severe chronic graft-versus-host disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

* Active, clinically diagnosed, moderate or severe cGVHD per NIH Consensus Criteria
* Underwent allogeneic stem cell transplantation (allo-HCT)
* Karnofsky Performance Status score ≥ 60%.
* Evidence of myeloid and platelet engraftment.
* Willingness to avoid pregnancy or fathering children based on protocol-defined criteria.

Exclusion Criteria:

* Has received more than 3 days/72 hours of systemic corticosteroid treatment for cGVHD.
* Has received any other systemic treatment for cGVHD, including extracorporeal photopheresis (ECP).
* Prior treatment with a Janus kinase (JAK) inhibitor for acute GVHD, unless the participant achieved complete or partial response and has been off JAK inhibitor treatment for at least 8 weeks before randomization.
* cGVHD occurring after a nonscheduled donor lymphocyte infusion (DLI) administered for pre-emptive treatment of malignancy recurrence.
* Evidence of relapsed primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, MD, Study Director — Incyte Corporation
Locations (133):
- United States (39):
  - University of Arizona Cancer Center - Out Pt., Tucson, Arizona
  - University of Arkansas For Medical Sciences - Winthrop P Rockefeller Cancer Institute, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Medical Center, Moores Cancer Center, La Jolla, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta University - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Cancer Specialists, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Hospital - Oncology Specislists Sc, Park Ridge, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital Authority, Westwood, Kansas
  - Tulane University, New Orleans, Louisiana
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester, James P. Wilmot Cancer Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tri Star Bone Marrow Transplant, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - St David'S South Austin Medical Center, Austin, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Ordensklinikum Linz Gmbh Elisabethinen, Linz, Austria
- Belgium (7):
  - Zna Stuivenberg, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
  - CENTRE HOSPITALIER UNIVERSITAIRE DE LIï¿½GE - SART TILMAN, Liège
  - AZ DELTA, Roeselare
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - University Health Network, Toronto, Ontario
  - Hospital Maisonneuve Rosemont, Montreal, Quebec
  - Saskatchewan Cancer, Saskatoon, Saskatchewan
- The Finsen Centre National Hospital, Copenhagen, Denmark
- Turku University Hospital, Turku, Finland
- France (10):
  - Chu Amiens Picardie - Hopital Sud, Amiens
  - Centre Hospitalier D'Angers, Angers
  - Chu de Grenoble - Hopital Albert Michallon, Grenoble
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Chu de Nice - Hospital L Archet, Nice
  - Chu de Rennes - Hospital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Chru Hopitaux de Tours Hospital Bretonneau, Tours
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (16):
  - Charite Berlin, Berlin
  - Universitatsklinikum Bonn Aoer, Bonn
  - Universitatsklinikum Koln, Cologne
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - Universitaetsklinikum Erlangen - Medizinische Klinik 5, Erlangen
  - Universitatsklinikum Essen, Essen
  - UNIVERSITï¿½TSKLINIKUM HALLE (SAALE), Halle
  - University Medical Centre Hamburg-Eppendorf Centre of Oncology, Hamburg
  - Universitaetsklinikum Jena, Jena
  - Selbststandige Abteilung Fur Hamatologie Und Internistische Onkologie, Leipzig
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - University Hospital Mannheim, Mannheim
  - Iii Medizinische Klinik Und Poliklinik Klinikum Rechts Der Isar Technische Universitat Munchen, Munich
  - Universitatsklinikum Munster, Münster
  - Universitaetsmedizin Rostock, Rostock
  - Universitaetsklinikum in Tubingen, Tübingen
- Greece (2):
  - University Hospital of West Attica - Attikon, Chaïdári
  - General Hospital of Thessaloniki G. Papanikolaou, Thessaloniki
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petach Tiqwa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (19):
  - CLINICA DI EMATOLOGIA, UNIVERSITï¿½ POLITECNICA DELLE MARCHE, Ancona
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo
  - L AZIENDA OSPEDALIERO-UNIVERSITARIA DI BOLOGNA POLICLINICO S. ORSOLA ï¿½ MALPIGHI, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Azienda Policlinico Vittorio Emanuele, Catania
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - A.O.U. Di Modena - Policlinico, Modena
  - A.O.U. Federico Ii, Napoli
  - Azienda Ospedaliera Ospedali Riuniti "Villa Sofia - Cervello", Palermo
  - Comitato Di Bioetica Della Fondazione Irccs Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli Ospedali Riuniti, Reggio Calabria
  - Universita Degli Studi Di Roma La Sapienza - Umberto I Policlinico Di Roma - Centro Di Ematologia, Roma
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Roma
  - Irrcs Instituto Clinico Humanitas, Rozzano
  - I.R.C.C.S. Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero Universitaria Citta Della Salute E Della Scienza, Torino
  - Azienda Ospedaliero-Universitaria Santa Maria Della Misericordia, Udine
  - Centro Ricerche Cliniche Di Verona (Crc), Verona
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii Im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy Oddzial W Gliwi, Gliwice
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
  - Mtz Clinical Research Sp. Zo.O., Warsaw
- Spain (14):
  - Institut Catala D Oncologia, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Ico Institut Catala D Oncologia, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Son Espases University Hospital, Palma
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Y Politcnico de La Fe, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Karolinska University Hospital Huddinge, Huddinge
  - Skane University Hospital Lund, Lund
- Universitatsspital Zurich, Zurich, Switzerland
- United Kingdom (8):
  - Bristol Haematology & Oncology Centre, Bristol
  - University Hospital of Wales, Cardiff
  - Barts Health Nhs Trust - St Bartholomews Hospital, London
  - King'S College Hospital (Nhs Foundation), London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton
  - St. George'S University Hospitals Nhs Foundation Trust, Tooting

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 65 study centers in Austria, Belgium, Canada, Denmark, Germany, Greece, Israel, Italy, Poland, Spain, Switzerland, United Kingdom, and the United States.
Groups:
- Part 1: Itacitinib 200 mg QD + CS: Participants were treated with oral itacitinib 200 milligrams (mg) once daily (QD) + corticosteroids (CS) for a maximum of 36 months. CS were given at a starting dose of 0.5 to 1.0 mg/kilogram (kg) QD (prednisone or methylprednisolone equivalent to prednisone dose). Itacitinib treatment was to continue until treatment failure (chronic graft-versus-host disease [cGVHD] progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months.
- Part 1: Itacitinib 300 mg QD + CS: Participants were treated with oral itacitinib 300 mg QD + CS for a maximum of 36 months. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). Itacitinib treatment was to continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months.
- Part 1 Expansion: Itacitinib 300 mg QD + CS: Participants were treated with oral itacitinib 300 mg QD + CS. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). Itacitinib treatment was to continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months.
- Part 1 Expansion: Itacitinib 400 mg QD + CS: Participants were treated with oral itacitinib 400 mg QD + CS. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). Itacitinib treatment was to continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months.
- Part 1 Expansion: Itacitinib 300 mg BID + CS: Participants were treated with oral itacitinib 300 mg twice daily (BID) + CS. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). The itacitanib dose could have been decreased to 200 mg BID if a boundary was reached during safety run-in. This treatment group was discontinued due to concern of a potential increase in relapse rate. Participants in this treatment group who were ongoing were allowed to reduce to 400 mg QD plus CS. Itacitinib treatment was to continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months.
- Part 1 Expansion: CS Monotherapy: Participants were treated with CS alone. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). Treatment was to continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months.
Period: Part 1
Arm/Group | Part 1: Itacitinib 200 mg QD + CS | Part 1: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Started | 11 | 10 | 0 | 0 | 0 | 0
Completed | 6 | 5 | 0 | 0 | 0 | 0
Not Completed | 5 | 5 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 2 | 0 | 0 | 0 | 0
Period: Part 1 Expansion
Arm/Group | Part 1: Itacitinib 200 mg QD + CS | Part 1: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Started | 0 | 0 | 35 | 39 | 29 | 36
Completed | 0 | 0 | 3 | 2 | 1 | 1
Not Completed | 0 | 0 | 32 | 37 | 28 | 35
Not completed — Death | 0 | 0 | 9 | 8 | 4 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 4 | 3 | 2 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 17 | 20 | 20 | 23
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 4 | 2 | 3
Not completed — Discontinued Treatment and Terminated CS Tapering | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression; cGVHD Flare | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Itacitinib 200 mg QD + CS | Part 1: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy | Total
Number analyzed (Participants) | 11 | 10 | 35 | 39 | 29 | 36 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (7.07) | 58.4 (15.08) | 53.6 (14.01) | 52.6 (13.79) | 52.6 (12.86) | 55.7 (13.32) | 54.2 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 17 | 16 | 14 | 19 | 72
  Male | 8 | 7 | 18 | 23 | 15 | 17 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 11 | 8 | 31 | 36 | 27 | 34 | 147
  Black/African-American | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Asian | 0 | 1 | 1 | 3 | 2 | 1 | 8
  Captured as "Other" in Database | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6 | 8 | 1 | 5 | 26
  Not Hispanic or Latino | 6 | 8 | 25 | 26 | 19 | 29 | 113
  Not Reported | 1 | 0 | 2 | 2 | 4 | 2 | 11
  Unknown | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Captured as "Other" in Database | 0 | 0 | 0 | 2 | 4 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any protocol-defined toxicity with onset up to and including Day 28, except those with a clear alternative explanation. Participants who received at least 21 of 28 doses of study drug at the level assigned or had a DLT were considered evaluable for determining tolerability of the dose. Participants who did not achieve this duration of exposure and did not have a DLT were to be replaced for purposes of toxicity identification.
Time Frame: up to Day 28
Population: Safety Analysis Set: all enrolled/randomized participants who received at least 1 dose of study drug and/or reference therapy. Treatment groups for this population were determined according to the actual treatment the participant received regardless of assigned study drug treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Itacitinib 200 mg QD + CS | Part 1: Itacitinib 300 mg QD + CS
Number analyzed (Participants) | 11 | 10
Participants | 0 | 1

2. Primary Outcome: Part 1 Expansion: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: until at least 30 days after the last dose of study treatment (up to 1103 days)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 39 | 29 | 36
Participants | 34 | 38 | 28 | 32

3. Primary Outcome: Part 2: Response Rate at Month 6
Description: Response rate was defined as the percentage of participants that had complete response (CR) or partial response (PR), per National Institutes of Health (NIH) Consensus Criteria, as determined by the investigator, within 14 days of the post-Baseline visit date until new anti-GVHD therapy or overall response-progression or relapse/progression of underlying disease. CR was defined as the complete resolution of all signs and symptoms of cGvHD in all evaluable organs. PR was defined as an improvement in at least one organ without progression in other organs.
Time Frame: Month 6
Population: Part 2 was not enrolled because the benefit:risk ratio did not support moving the combination of itacitinib with CS to a later phase of development in first-line cGVHD.
Groups:
- Part 2: Itacitinib QD + CS: Participants were to be treated with oral itacitinib QD at the recommended Part 2 dose + CS. CS were to be given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose).
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

4. Secondary Outcome: Part 1 Expansion: Response Rate at Months 3 and 6
Description: Response rate was defined as the percentage of participants that had CR or PR, per NIH Consensus Criteria, as determined by the investigator, within 14 days of the post-Baseline visit date until new anti-GVHD therapy or overall response-progression or relapse/progression of underlying disease. CR was defined as the complete resolution of all signs and symptoms of cGvHD in all evaluable organs. PR was defined as an improvement in at least one organ without progression in other organs.
Time Frame: Months 3 and 6
Population: Safety Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 39 | 29 | 36
percentage of participants
  Month 3 | 60.0 [42.1 to 76.1] | 69.2 [52.4 to 83.0] | 58.6 [38.9 to 76.5] | 50.0 [32.9 to 67.1]
  Month 6 | 42.9 [26.3 to 60.6] | 53.8 [37.2 to 69.9] | 34.5 [17.9 to 54.3] | 36.1 [20.8 to 53.8]

5. Secondary Outcome: Parts 1 and 1 Expansion: Cmax of Itacitinib
Description: Cmax was defined as the maximum observed concentration of itacitinib.
Time Frame: Days 1, 7, and 28: predose and 1, 2, and 5 hours post-dose
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of study drug and/or reference therapy and provided at least 1 corresponding post-dose plasma sample (1 PK measurement). Because Part I and Part I Expansion were both randomized, open label, and had a parallel design with the same participant population criteria, as pre-specified, the PK data for identical doses/frequency of dosing were grouped for analysis (rather than conducting analysis by treatment arm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per Liter (nmol/L)
Groups:
- Parts 1 and 1 Expansion: 100 mg QD + CS: For toxicity management purposes and/or due to coadministration of strong CYP3A4 inhibitors, participants who received a starting dose of itacitinib 200 mg or 300 mg QD + CS in Part 1 and a starting dose of itacitinib 300 mg or 400 mg QD + CS in Part 1 Expansion had first or second dose reductions to itacitinib 100 mg QD + CS and/or dose interruptions.
- Parts 1 and 1 Expansion: Itacitinib 200 mg QD + CS: Participants were treated with a starting dose of oral itacitinib 200 mg QD + CS in Part 1 or had a dose reduction to oral itacitinib 200 mg QC + CS in Part 1 or Part 1 Expansion. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). For toxicity management purposes and/or due to coadministration of strong CYP3A4 inhibitors, participants who received a starting dose of itacitinib 300 mg QD + CS in Part 1 and a starting dose of itacitinib 300 mg or 400 mg QD + CS in Part 1 Expansion had first or second dose reductions to itacitinib 200 mg QD + CS and/or dose interruptions.
- Parts 1 and 1 Expansion: Itacitinib 300 mg QD + CS: Participants were treated with a starting dose of oral itacitinib 300 mg QD + CS in Part 1 or Part 1 Expansion or had a dose reduction to oral itacitinib 300 mg QC + CS in Part 1 Expansion. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). Itacitinib treatment was to continue until treatment failure (chronic graft-versus-host disease [cGVHD] progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months. For toxicity management purposes and/or due to coadministration of strong CYP3A4 inhibitors, participants who received a starting dose of itacitinib 400 mg QD + CS in Part 1 Expansion had a dose reduction to itacitinib 300 mg QD + CS and/or dose interruptions.
- Part 1 Expansion: Itacitinib 100 mg BID + CS: For toxicity management purposes and/or due to coadministration of strong CYP3A4 inhibitors, participants who received a starting dose of itacitinib 300 mg BID + CS in Part 1 Expansion had first or second dose reductions to itacitinib 100 mg BID + CS and/or dose interruptions.
- Part 1 Expansion: Itacitinib 200 mg BID + CS: Participants were treated with a starting dose of oral itacitinib 300 mg BID + CS in Part 1 Expansion and had their dose decreased to itacitinib 200 mg BID + CS because a boundary was reached during safety run-in or for toxicity management purposes and/or due to coadministration of strong CYP3A4 inhibitors. CS were given at a starting dose of 0.5 to 1.0 mg/kg QD (prednisone or methylprednisolone equivalent to prednisone dose). Itacitinib treatment was to continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months. For toxicity management purposes and/or due to coadministration of strong CYP3A4 inhibitors, participants who received a starting dose of itacitinib 300 mg BID + CS in Part 1 Expansion had a dose reduction to itacitinib 200 mg BID + CS and/or dose interruptions.
Arm/Group | Parts 1 and 1 Expansion: 100 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 200 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 100 mg BID + CS | Part 1 Expansion: Itacitinib 200 mg BID + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS
Number analyzed (Participants) | 3 | 27 | 35 | 26 | 3 | 14 | 16
nanomoles per Liter (nmol/L)
  Day 1: number analyzed (Participants) | 1 | 23 | 35 | 26 | 0 | 12 | 16
  Day 1 | 201 (NA) — SD cannot be reported for a single participant. | 655 (82.9) | 1050 (87.3) | 951 (68.0) |  | 769 (118) | 736 (79.1)
  Day 7: number analyzed (Participants) | 1 | 27 | 32 | 26 | 0 | 14 | 12
  Day 7 | 191 (NA) — SD cannot be reported for a single participant. | 1070 (88.9) | 1580 (125) | 1190 (103) |  | 1520 (73.0) | 1110 (66.2)
  Day 28: number analyzed (Participants) | 3 | 26 | 27 | 21 | 3 | 8 | 10
  Day 28 | 486 (140) | 1460 (67.3) | 1290 (248) | 1350 (72.2) | 1350 (29.4) | 2040 (62.6) | 1580 (51.4)

6. Secondary Outcome: Parts 1 and 1 Expansion: Ctau of Itacitinib
Description: Ctau was defined as the trough concentration of itacitinib over the dose interval. For pharmacokinetic steady state Day 7 and Day 28, for the calculation of NCA exposure estimates (as more than 3 PK data points are necessary for the estimation beyond Cmax) it was assumed, that PK concentration returns to the predose value (at 12 hours post-dose for BID dosing; at 24 hours post-dose for QD dosing). Predose PK samples were transposed to 24 hours post-dose for QD administration and to 12 hours post-dose for BID administration to allow the steady-state NCA PK estimates on Day 7 and Day 28.
Time Frame: Day 1: predose, and 1, 2, and 5 hours post-dose. Days 7 and 28: predose, and 1, 2, 5, 12 (for BID dosing), and 24 hours post-dose (for QD dosing)
Population: PK Evaluable Population. Because Part I and Part I Expansion were both randomized, open label, and had a parallel design with the same participant population criteria, as pre-specified, the PK data for identical doses/frequency of dosing were grouped for analysis (rather than conducting analysis by treatment arm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Parts 1 and 1 Expansion: 100 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 200 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 100 mg BID + CS | Part 1 Expansion: Itacitinib 200 mg BID + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS
Number analyzed (Participants) | 3 | 27 | 35 | 26 | 3 | 14 | 16
nmol/L
  Day 1: number analyzed (Participants) | 1 | 23 | 35 | 26 | 0 | 12 | 16
  Day 1 | NA (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Ctau (as more than 3 PK data points are necessary beyond Cmax). | NA (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Ctau (as more than 3 PK data points are necessary beyond Cmax). | 0.153 (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Ctau (as more than 3 PK data points are necessary beyond Cmax). Of the total participants analyzed, only 1 participant had a PK profile that allowed for the NCA estimate of the parameter. Thus, the calculation of the SD was not possible. | 135 (197) |  | 7.54 (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Ctau (as more than 3 PK data points are necessary beyond Cmax). Of the total participants analyzed, only 1 participant had a PK profile that allowed for the NCA estimate of the parameter. Thus, the calculation of the SD was not possible. | NA (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Ctau (as more than 3 PK data points are necessary beyond Cmax).
  Day 7: number analyzed (Participants) | 1 | 27 | 31 | 24 | 0 | 14 | 12
  Day 7 | 0.298 (NA) — SD cannot be reported for a single participant. | 53.6 (218) | 52.2 (425) | 33.5 (118) |  | 483 (175) | 127 (177)
  Day 28: number analyzed (Participants) | 3 | 26 | 26 | 20 | 3 | 8 | 10
  Day 28 | 10.4 (4440) | 68.0 (314) | 42.2 (182) | 29.7 (152) | 392 (85.6) | 460 (123) | 195 (116)

7. Secondary Outcome: Parts 1 and 1 Expansion: Tmax of Itacitinib
Description: tmax was defined as the time to the maximum concentration of itacitinib. For pharmacokinetic steady state Day 7 and Day 28, for the calculation of NCA exposure estimates (as more than 3 PK data points are necessary for the estimation beyond Cmax) it was assumed, that PK concentration returns to the predose value (at 12 hours post-dose for BID dosing; at 24 hours post-dose for QD dosing). Predose PK samples were transposed to 24 hours post-dose for QD administration and to 12 hours post-dose for BID administration to allow the steady-state NCA PK estimates on Day 7 and Day 28.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Parts 1 and 1 Expansion: 100 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 200 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 100 mg BID + CS | Part 1 Expansion: Itacitinib 200 mg BID + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS
Number analyzed (Participants) | 3 | 27 | 35 | 26 | 3 | 14 | 16
hours
  Day 1: number analyzed (Participants) | 1 | 23 | 35 | 26 | 0 | 12 | 16
  Day 1 | 1.0 [1.0 to 1.0] | 2.1 [0.9 to 4.8] | 2.1 [0.8 to 5.0] | 2.0 [0.0 to 5.0] |  | 2.0 [1.0 to 5.0] | 2.4 [1.0 to 5.0]
  Day 7: number analyzed (Participants) | 1 | 27 | 32 | 26 | 0 | 14 | 12
  Day 7 | 1.0 [1.0 to 1.0] | 2.1 [0.0 to 5.0] | 2.0 [1.0 to 13.4] | 2.0 [1.0 to 5.2] |  | 1.9 [0.0 to 10.7] | 2.0 [0.9 to 5.0]
  Day 28: number analyzed (Participants) | 3 | 26 | 27 | 21 | 3 | 8 | 10
  Day 28 | 4.0 [1.0 to 4.8] | 3.1 [0.8 to 12.0] | 2.0 [0.0 to 16.9] | 2.1 [0.9 to 5.0] | 2.0 [2.0 to 2.2] | 2.3 [2.0 to 5.6] | 2.0 [1.0 to 5.0]

8. Secondary Outcome: Parts 1 and 1 Expansion: Cl/F of Itacitinib
Description: Cl/F was defined as the apparent oral dose clearance of itacitinib. For pharmacokinetic steady state Day 7 and Day 28, for the calculation of NCA exposure estimates (as more than 3 PK data points are necessary for the estimation beyond Cmax) it was assumed, that PK concentration returns to the predose value (at 12 hours post-dose for BID dosing; at 24 hours post-dose for QD dosing). Predose PK samples were transposed to 24 hours post-dose for QD administration and to 12 hours post-dose for BID administration to allow the steady-state NCA PK estimates on Day 7 and Day 28.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Parts 1 and 1 Expansion: 100 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 200 mg QD + CS | Parts 1 and 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 100 mg BID + CS | Part 1 Expansion: Itacitinib 200 mg BID + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS
Number analyzed (Participants) | 3 | 27 | 35 | 26 | 3 | 14 | 16
Liters per hour
  Day 1: number analyzed (Participants) | 1 | 23 | 35 | 26 | 0 | 12 | 16
  Day 1 | NA (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Cl/F (as more than 3 PK data points are necessary beyond Cmax). | NA (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Cl/F (as more than 3 PK data points are necessary beyond Cmax). | 258 (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Cl/F (as more than 3 PK data points are necessary beyond Cmax). Of the total participants analyzed, only 1 participant had a PK profile that allowed for the NCA estimate of the parameter. Thus, the calculation of the SD was not possible. | 41.2 (130) |  | 640 (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Cl/F (as more than 3 PK data points are necessary beyond Cmax). Of the total participants analyzed, only 1 participant had a PK profile that allowed for the NCA estimate of the parameter. Thus, the calculation of the SD was not possible. | NA (NA) — The absence of terminal PK measurements at baseline visits for the timepoint beyond 6 hours did not allow for precise and reasonable NCA estimates related to Cl/F (as more than 3 PK data points are necessary beyond Cmax).
  Day 7: number analyzed (Participants) | 1 | 27 | 31 | 24 | 0 | 14 | 12
  Day 7 | 224 (NA) — SD cannot be reported for a single participant. | 43.0 (105) | 48.9 (159) | 85.9 (90.7) |  | 31.8 (82.9) | 94.4 (61.3)
  Day 28: number analyzed (Participants) | 3 | 26 | 26 | 20 | 3 | 8 | 10
  Day 28 | 47.7 (211) | 30.0 (96.9) | 54.8 (189) | 81.0 (65.1) | 20.2 (54.2) | 26.9 (75.5) | 67.5 (62.1)

9. Secondary Outcome: Part 2: Cmax of Itacitinib
Description: Cmax was defined as the maximum observed concentration of itacitinib.
Time Frame: Days 1, 7, and 28: predose and 1, 2, and 5 hours post-dose
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

10. Secondary Outcome: Part 2: Cmin of Itacitinib
Description: Cmin was defined as the minimum observed plasma or serum concentration of itacitinib over the dose interval.
Time Frame: Days 1, 7, and 28: predose and 1, 2, and 5 hours post-dose
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

11. Secondary Outcome: Part 2: Tmax of Itacitinib
Description: tmax was defined as the time to the maximum concentration of itacitinib.
Time Frame: Days 1, 7, and 28: predose and 1, 2, and 5 hours post-dose
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

12. Secondary Outcome: Part 2: AUC0-t of Itacitinib
Description: AUC0-t was defined as the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Time Frame: Days 1, 7, and 28: predose and 1, 2, and 5 hours post-dose
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

13. Secondary Outcome: Part 2: Cl/F of Itacitinib
Description: Cl/F was defined as the apparent oral dose clearance of itacitinib.
Time Frame: Days 1, 7, and 28: predose and 1, 2, and 5 hours post-dose
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

14. Secondary Outcome: Part 1: Response Rate at Months 3, 6, and 12
Description: as for outcome 4
Time Frame: Months 3, 6, and 12
Population: Safety Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Itacitinib 200 mg QD + CS | Part 1: Itacitinib 300 mg QD + CS
Number analyzed (Participants) | 11 | 10
percentage of participants
  Month 3 | 63.6 [30.8 to 89.1] | 50.0 [18.7 to 81.3]
  Month 6 | 36.4 [10.9 to 69.2] | 50.0 [18.7 to 81.3]
  Month 12 | 18.2 [2.3 to 51.8] | 20.0 [2.5 to 55.6]

15. Secondary Outcome: Part 1 Expansion: Response Rate at Month 12
Description: as for outcome 4
Time Frame: Month 12
Population: Safety Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 39 | 29 | 36
percentage of participants | 22.9 [10.4 to 40.1] | 41.0 [25.6 to 57.9] | 24.1 [10.3 to 43.5] | 19.4 [8.2 to 36.0]

16. Secondary Outcome: Part 1 Expansion: Time to Response
Description: Time to response was defined as the interval between randomization and the first response (CR or PR) before initiation of new therapy. CR was defined as the complete resolution of all signs and symptoms of cGvHD in all evaluable organs. PR was defined as an improvement in at least one organ without progression in other organs.
Time Frame: up to Month 12
Population: Safety Analysis Set. Participants with a first response of CR or PR up to 12 months, until initiation of new anti-GVHD therapy, relapse of underlying malignancy, or overall response of progression or death were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 31 | 31 | 25 | 26
days | 16.0 [12 to 120] | 16.0 [12 to 86] | 16.0 [13 to 145] | 16.0 [13 to 88]

17. Secondary Outcome: Part 1 Expansion: Duration of Response
Description: Duration to response was defined as the interval between the first response and cGVHD progression, death, or the initiation of a new systemic cGVHD therapy.
Time Frame: up to 24 months
Population: Safety Analysis Set. Participants with a first response of CR or PR up to 12 months, until initiation of new anti-GVHD therapy, relapse of underlying malignancy, or overall response of progression or death were analyzed. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 31 | 31 | 25 | 26
days | 581.0 [147.0 to 807.0] | NA [306.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died or initiated new systemic cGVHD therapy. | 512.0 [161.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died or initiated new systemic cGVHD therapy. | 197.0 [103.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died or initiated new systemic cGVHD therapy.

18. Secondary Outcome: Part 1 Expansion: Overall Survival
Description: Overall survival was defined as the interval between the date of randomization and the date of death due to any cause.
Time Frame: up to 36 months
Population: Safety Analysis Set. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 39 | 29 | 36
days | NA [694.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants died.

19. Secondary Outcome: Part 1 Expansion: Nonrelapse Mortality (NRM) Rate
Description: NRM was defined as the percentage of participants who died due to causes other than a relapse of their primary hematologic disease.
Time Frame: up to 24 months
Population: Safety Analysis Set. Participants who did not die due to malignancy relapse were analyzed. The 95% confidence interval was calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 37 | 28 | 35
percentage of participants | 25.7 [12.5 to 43.3] | 15.4 [6.2 to 32.0] | 10.3 [2.3 to 28.2] | 11.1 [3.2 to 26.7]

20. Secondary Outcome: Part 1 Expansion: Percentage of Participants With a ≥50% Reduction in Daily Corticosteroid Dose at Day 180 From the Corticosteroid Dose on Day 1
Description: The corticosteroid dose at Day 180 was compared to the corticosteroid dose on Day 1 to assess reduction.
Time Frame: Day 1; Day 180
Population: Safety Analysis Set. Only those participants ongoing in the study at Day 180 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 21 | 27 | 17 | 18
percentage of participants | 90.5 | 100.0 | 100.0 | 100.0

21. Secondary Outcome: Part 1 Expansion: Percentage of Participants Successfully Tapered Off All Corticosteroids at Day 180
Description: The percentage of participants who were not taking any corticosteroids at Day 180 was assessed.
Time Frame: Day 180
Population: Safety Analysis Set. Only those participants ongoing in the study at Day 180 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 21 | 27 | 17 | 18
percentage of participants | 52.4 | 66.7 | 47.1 | 44.4

22. Secondary Outcome: Part 1 Expansion: Relapse Rate of Malignant and Nonmalignant Hematologic Diseases
Description: The relapse rate was defined as the percentage of participants whose underlying disease relapsed at any time during the course of the study.
Time Frame: up to 1073 days
Population: Safety Analysis Set. The 95% confidence interval was calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 39 | 29 | 36
percentage of participants | 5.7 [0.7 to 19.2] | 7.7 [1.6 to 20.9] | 13.8 [3.9 to 31.7] | 2.8 [0.1 to 14.5]

23. Secondary Outcome: Part 1 Expansion: Time to Primary Hematologic Disease Relapse
Description: Time to primary hematologic disease relapse was defined as the interval between the date of randomization and the date of relapse.
Time Frame: up to 24 months
Population: Safety Analysis Set, including censored participants. Censored participants didn't have an event of relapse at any time up to the last assessment date. Participants who didn't have an event of hematologic disease relapse were censored at the time of the last assessment. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: CS Monotherapy
Number analyzed (Participants) | 35 | 39 | 29 | 36
days | NA [NA to NA] — Too few participants had an event of relapse for a meaningful median/95% confidence interval to be calculated; thus, the Kaplan-Meier estimator cannot provide a valid estimate. | NA [NA to NA] — Too few participants had an event of relapse for a meaningful median/95% confidence interval to be calculated; thus, the Kaplan-Meier estimator cannot provide a valid estimate. | NA [NA to NA] — Too few participants had an event of relapse for a meaningful median/95% confidence interval to be calculated; thus, the Kaplan-Meier estimator cannot provide a valid estimate. | NA [NA to NA] — Too few participants had an event of relapse for a meaningful median/95% confidence interval to be calculated; thus, the Kaplan-Meier estimator cannot provide a valid estimate.

24. Secondary Outcome: Part 2: Change From Baseline in Lee cGVHD Symptom Scale (LLS) Scores
Description: The LSS consists of 30 items in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological). It was to be used to assess patient-reported changes in health status, symptoms, and well being.
Time Frame: Baseline; End of Treatment in Phase 2
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 2: Change From Baseline in Quality of Life-Short Form-36 Version 2 (QOL-SF-36 v2) Scores
Description: The QOL-SF-36 v2 is 36-item scale that captures changes in health status during the course of treatment. The SF-36 assesses 8 health concepts related to limitations in physical activities, social activities, bodily pain, general mental and physical health, and vitality. It was to be used to assess patient-reported changes in health status, symptoms, and well being.
Time Frame: Baseline; End of Treatment in Phase 2
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 2: Change From Baseline in EQ-5D-3L Scores
Description: The EQ-5D-3L is a descriptive classification consisting of 5 dimensions of health: mobility, self-care, usual activities, anxiety/depression, and pain/discomfort. It was to be used to assess patient-reported changes in health status, symptoms, and well being.
Time Frame: Baseline; End of Treatment in Phase 2
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 2: Change From Baseline in Patient Global Impression of Change (PGIC) Responses
Description: The PGIC is 1 question that captures the overall change in symptoms over the course of treatment. It was to be used to assess patient-reported changes in health status, symptoms, and well being.
Time Frame: Baseline; End of Treatment in Phase 2
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 2: Change From Baseline in Patient Global Impression of Severity (PGIS) Responses
Description: The PGIS is 1 question that captures the overall change in the severity of symptoms over the previous week. It was to be used to assess patient-reported changes in health status, symptoms, and well being.
Time Frame: Baseline; End of Treatment in Phase 2
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

29. Secondary Outcome: Part 2: Response Rate at Months 3 and 12
Description: as for outcome 4
Time Frame: Months 3 and 12
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

30. Secondary Outcome: Part 2: Duration of Response
Description: as for outcome 17
Time Frame: up to 24 months
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

31. Secondary Outcome: Part 2: Overall Survival
Description: Overall survival was defined as the interval between the date of randomization and the date of death due to any cause.
Time Frame: up to 36 months
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 2: NRM Rate
Description: as for outcome 19
Time Frame: up to 24 months
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

33. Secondary Outcome: Part 2: Percentage of Participants With a ≥50% Reduction in Daily Corticosteroid Dose at Day 180 From the Corticosteroid Dose on Day 1
Description: The corticosteroid dose at Day 180 was compared to the corticosteroid dose on Day 1 to assess reduction.
Time Frame: Day 1; Day 180
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

34. Secondary Outcome: Part 2: Percentage of Participants Successfully Tapered Off All Corticosteroids at Day 180
Description: The percentage of participants who were not taking any corticosteroids at Day 180 was assessed.
Time Frame: Day 180
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 2: Relapse Rate of Malignant and Nonmalignant Hematologic Diseases
Description: The relapse rate was defined as the defined as the percentage of participants whose underlying disease relapsed at any time during the course of the study.
Time Frame: up to 24 months
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 2: Time to Primary Hematologic Disease Relapse
Description: as for outcome 23
Time Frame: up to 24 months
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

37. Secondary Outcome: Part 2: Number of Participants With Any TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 30 days after the last dose in Phase 2
Population: as for outcome 3
Arm/Group | Part 2: Itacitinib QD + CS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: until at least 30 days after the last dose of study treatment (up to 1103 days)
Description: Treatment-emergent adverse events (TEAEs), defined as any AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug, have been reported. As pre-specified in the SAP, the overall summary of AEs by treatment group included the number of participants with itacitinib dose reductions due to AEs or concomitant strong CYP3A4 inhibitors. The SAP defines "treatment groups" as those to which participants were originally randomized.
Groups:
- Part 1 Expansion: Total: Participants received 300 mg QD, 400 mg QD, or 300 mg BID itacitinib plus corticosteroids.
Arm/Group | Part 1: Itacitinib 200 mg QD + CS | Part 1: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg QD + CS | Part 1 Expansion: Itacitinib 400 mg QD + CS | Part 1 Expansion: Itacitinib 300 mg BID + CS | Part 1 Expansion: Total | Part 1 Expansion: CS Monotherapy
All-Cause Mortality (participants affected / at risk) | 2/11 | 3/10 | 9/35 | 8/39 | 4/29 | 21/103 | 5/36
Serious Adverse Events (participants affected / at risk) | 6/11 | 5/10 | 18/35 | 22/39 | 12/29 | 52/103 | 9/36
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10 | 33/35 | 37/39 | 27/29 | 97/103 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Itacitinib 200 mg QD + CS (N=11) | Part 1: Itacitinib 300 mg QD + CS (N=10) | Part 1 Expansion: Itacitinib 300 mg QD + CS (N=35) | Part 1 Expansion: Itacitinib 400 mg QD + CS (N=39) | Part 1 Expansion: Itacitinib 300 mg BID + CS (N=29) | Part 1 Expansion: Total (N=103) | Part 1 Expansion: CS Monotherapy (N=36)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis obliterans syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 6 (6) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clostridial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (3) | 5 (5) | 2 (2) | 9 (10) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salmonella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Systemic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Itacitinib 200 mg QD + CS (N=11) | Part 1: Itacitinib 300 mg QD + CS (N=10) | Part 1 Expansion: Itacitinib 300 mg QD + CS (N=35) | Part 1 Expansion: Itacitinib 400 mg QD + CS (N=39) | Part 1 Expansion: Itacitinib 300 mg BID + CS (N=29) | Part 1 Expansion: Total (N=103) | Part 1 Expansion: CS Monotherapy (N=36)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 1 (2) | 7 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 5 (7) | 6 (14) | 6 (10) | 17 (31) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 14 (18) | 9 (13) | 10 (12) | 33 (43) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (4) | 3 (4) | 9 (11) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 0 (0) | 3 (5) | 4 (6) | 2 (4) | 9 (15) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (2) | 2 (2) | 7 (9) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 7 (7) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Blood cholesterol increased (Investigations) | 3 (3) | 2 (2) | 3 (3) | 4 (5) | 4 (4) | 11 (12) | 1 (2)
Blood creatinine increased (Investigations) | 3 (6) | 2 (2) | 3 (3) | 4 (7) | 3 (5) | 10 (15) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 4 (4) | 14 (14) | 5 (5)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 7 (7) | 2 (2) | 13 (13) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 6 (6) | 3 (4)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2) | 1 (1) | 3 (6) | 8 (14) | 4 (5) | 15 (25) | 3 (6)
Cytomegalovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 9 (10) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 6 (6) | 4 (6) | 6 (9) | 16 (21) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 7 (7) | 2 (2)
Drug level increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 6 (7) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 2 (2) | 6 (7) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 5 (7) | 2 (2) | 1 (1) | 8 (10) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 5 (7) | 0 (0)
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 4 (6) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (3) | 1 (2) | 2 (2) | 4 (7) | 3 (3)
Fatigue (General disorders) | 4 (4) | 2 (3) | 6 (7) | 7 (8) | 4 (4) | 17 (19) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (2) | 6 (9) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (6) | 1 (1) | 9 (9) | 3 (4)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 4 (4) | 5 (5) | 4 (5) | 13 (14) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 3 (5) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (3) | 6 (6) | 7 (8) | 9 (10) | 22 (24) | 7 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 8 (9) | 3 (3) | 13 (14) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (3) | 0 (0) | 5 (7) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (6) | 6 (8) | 12 (16) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (9) | 2 (6) | 1 (3) | 8 (18) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (8) | 3 (5) | 3 (4) | 11 (17) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 2 (2) | 5 (7) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 8 (8) | 4 (5) | 15 (16) | 5 (5)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 6 (6) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 5 (5) | 4 (4) | 0 (0) | 9 (9) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 8 (10) | 5 (6) | 2 (2) | 15 (18) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (8) | 3 (11) | 3 (6) | 11 (25) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (5) | 0 (0)
Oedema (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 6 (6) | 5 (5) | 6 (7) | 17 (18) | 6 (6)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 5 (5) | 3 (3) | 6 (6) | 7 (7) | 9 (11) | 22 (24) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 4 (6) | 5 (6) | 6 (6) | 15 (18) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 4 (5) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 4 (5) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 6 (7) | 2 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 8 (9) | 7 (8) | 5 (5) | 20 (22) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 1 (1) | 5 (7) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 3 (4) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 6 (6) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (2) | 0 (0) | 5 (8) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Based on preliminary data, Part 2 did not enroll participants. All participants in Part 1 Expansion who were on treatment with either itacitinib 300 or 400 milligrams (mg) once daily (QD) and who were tolerating and continuing to receive benefit from itacitinib had the option to continue itacitinib treatment in the INCB 39110-801 (NCT04640025) roll-over study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03584516/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03584516/SAP_001.pdf